CLINICAL TRIAL: NCT02404870
Title: Acute Effects of Canagliflozin, a Sodium Glucose Co-Transporter 2 (SGLT2) Inhibitor on Bone Metabolism in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: 140195; 14-DK-0195
Record Dates: First submitted 2015-03-31; First posted 2015-04-01 (Estimated); Last update posted 2025-03-04 (Actual); Status verified 2025-03

CONDITIONS: Healthy Volunteers
Keywords: Diabetes; Phosphate; Fibroblast Growth Factor 23 (FGF23); Vitamin D; PTH
MeSH Terms: conditions — Diabetes Mellitus | interventions — Canagliflozin

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Admission 1 or 2 (Experimental): Canagliflozin
  Interventions: Drug: Canagliflozin
- Admission 2 or 1 (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Placebo — Placebo
  Arms: Admission 2 or 1
Drug: Canagliflozin — Canagliflozin is a new oral drug for the treatment of type 2 diabetes mellitus (T2DM), and is one of two recently FDA approved sodium glucose co-transporter 2 (SGLT2) inhibitors, which target renal glucose reabsorption and offer promising improvement in HbA1C.
  Arms: Admission 1 or 2

SUMMARY:
Background:

- Canagliflozin (sold as InvokanaTM) is a new medicine for diabetes. But it might increase the bone fracture risk in people with diabetes.

Objective:

- To see if Invokana has negative side effects on bone health.

Eligibility:

- Healthy men ages 18 45.

Design:

* Participants will be screened with a medical history, physical exam, and blood tests. A nutritionist will discuss their dietary history and the study dietary requirements. Participants will get a food diary to record what they eat and drink on 3 separate days.
* Participants will have a DEXA scan x-ray test of bone health. Participants will lie still on a table while a small camera passes over the body.
* Participants will have 2 stays in the clinic. They will be 1 week apart and each last 6 overnights starting on a Sunday.
* Before each stay, participants will:
* Pick up food each day for 7 days. They will get breakfast, lunch, dinner, and snacks. They must eat only the food provided during these times.
* Collect their urine twice.
* During the stays, participants will:
* Be evaluated by a doctor and have blood drawn.
* On each Monday, participants will:
* Skip breakfast
* At about 8 a.m. take a placebo pill in one stay, the study drug in the other stay.
* Drink 6 ounces of water every 2 hours for 4 hours.
* An intravenous (IV) catheter will be inserted into an arm. Blood will be drawn every 2 hours from 8 a.m. until noon.
* Get lunch.
* Have blood testing again at 8pm and midnight.
* Repeat the testing days 2 5.
* Have urine collected.

DETAILED DESCRIPTION:
Background

Canagliflozin is a new oral drug for the treatment of type 2 diabetes mellitus (T2DM), and is one of four recently FDA approved sodium glucose co-transporter 2 (SGLT2) inhibitors, which target renal glucose reabsorption and offer promising improvement in HbA1c. In the approval process, the FDA Advisory Committee reviewed data suggesting that canagliflozin increased the incidence of fractures. In addition, the drug induced changes in phosphate, bone resorption markers, parathyroid hormone (PTH) and vitamin D metabolism which might mediate the adverse changes in bone homeostasis. For a variety of reasons, the data on bone fracture risk are relatively limited. First, the drug s development program was focused primarily on demonstrating efficacy, and bone fractures were only one of many safety end-points which were monitored. Second, only a minority of patients (approximately 1%) experienced bone fractures in the course of the development program. Finally, there appears to be a lag time prior to the time increased bone resorption translates into a significant increase in the rate of bone fractures. We hypothesize that this class of drugs causes a cascade of hormonal changes induced by increased phosphorus reabsorption that leads to significant changes in fibroblast growth factor 23 (FGF23), PTH, and vitamin D metabolism which ultimately increase fracture risk.

Aim

The primary endpoint is to determine the effects of canagliflozin on bone health by evaluating changes in the area under the curve (AUC) of FGF23 during the first 24-72 hours. Secondary endpoints include the evaluation of canagliflozin on other biochemical parameters in the early phase (1 week) of drug administration during which we hypothesize a new steady state will be reached related to bone metabolism including PTH, 1,25 vitamin D, tubular reabsorption of phosphate (TRP), and carboxy-terminal telopeptide (CTX).

Methods

A randomized, blinded, placebo-controlled cross-over pilot study of healthy volunteers age 18 years and older with a BMI of 20 - 30 kg/m2.

Patients will be randomized to canagliflozin (300mg once daily) or placebo for 5 days and will be studied as inpatients (NIH Clinical Center metabolic unit). Serial blood and urine testing for 4 hours after daily drug administration and at 12 and 24 hours thereafter will be used to assess changes in the pre-specified endpoints. Each subject will be provided a diet containing fixed contents of phosphate, sodium, and calcium throughout the study, beginning 7 days prior to the administration of drug (or placebo).

ELIGIBILITY:
* INCLUSION CRITERIA:

We are targeting healthy men and women greater than or equal to 18 years old, inclusive of all races and ethnicity within a BMI of 20 30 kg/m(2). Specifically, we have defined healthy to mean: normal fasting glucose and hemoglobin A1c less than or equal to 6%, normal Hb, no glucosuria, normal renal function (based on normal serum creatinine + Cystatin C), urine albumin:creatinine ratio, protein:creatinine ratio, and GFR > 80 as calculated by the CKD-Epi equation and normal lab urinalysis.

EXCLUSION CRITERIA:

If you have any of the following health issues, you cannot participate in the study:

* Presence of heart disease, untreated high blood pressure (>140/90 mm Hg), orthostatic hypotension or symptomatic hypotension, cancer, diabetes, recurrent symptomatic hypoglycemia and /or history of recurrent genital or urinary tract infection, thyroid disease, or any other condition that affects bone health
* Past history of eating disorder or psychiatric disorders, including severe depression, anxiety, or psychosis or presently on treatment with medications for any of these conditions
* Taking certain medications, especially those that affect bone metabolism (e.g., high dose vitamin D [>1000 units daily] or calcium supplements [>800mg daily], high dose vitamin A [>20,000 units daily], phosphate binding antacids, calcitonin, calcitriol, growth hormone, or any anti-seizure medications for any reason including valproic acid, lamotrigine), certain medications for high blood pressure (diuretics), steroids including inhalers, diet/weight loss medications, or any other medications at the discretion of the principal investigator and/or study team
* Have started, increased or decreased calcium [>400mg daily] or vitamin D [>1000 units daily] supplements within 2 weeks of the study
* Dependence or regular use of alcohol (>2 drinks per day), tobacco (smoking or chewing), amphetamines, cocaine, heroin or marijuana over the past 6 months
* Volunteers will be excluded if they have abnormal blood concentrations of

  * inorganic phosphate level (less than or equal to 2.5 mg/dl or greater than or equal to 4.8 mg/dl),
  * parathyroid hormone (PTH) (less than or equal to 60 pg/ml),
  * creatinine (less than or equal to 1.5 mg/dl) or eGFR (< 80 ml/min/1.73sq.m),
  * fasting glucose (greater than or equal to 100 mg/dl),
  * hemoglobin (less than or equal to 11 g/dl),
  * liver function tests (more than twice normal),
  * testosterone (less than or equal to 260 ng/dl)
* Participation in a vigorous exercise program (>3h/day of vigorous activity)
* Consume more than 300 mg/day of caffeine (about two to three 8 fluid ounce servings)
* Have strict dietary concerns (e.g., vegan or kosher diet, multiple food allergies)
* Cannot commit to the research experience at the Clinical Research Center as required by the study timeline
* Have previous hypersensitivity reaction to canagliflozin (including but not limited to rash, raised red patches on your skin (hives), swelling of the face, lips, tongue, and throat that may cause difficulty in breathing or swallowing).
* Positive urine pregnancy test and/or planning to become pregnant during the course of the study.
* You are unwilling to use effective contraceptive methods for duration of study (hormonal or barrier.
* Irregular menstrual cycles

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2014-09-16 (Actual); Primary Completion 2019-05-01 (Actual); Study Completion 2019-09-03 (Actual)

PRIMARY OUTCOMES:
AUC of FGF23 | First 24-72 hours
  In this study, our primary endpoint is the area under the curve (AUC) for FGF23 for the 24-72 hours from the first day of administration of canagliflozin. The null hypothesis is that there will be no change in the mean 24-72 hours AUC of FGF23 after the treatment compared with the mean baseline value. We acknowledge that the magnitude and time course of changes (if any) in FGF23 are totally unknown.

SECONDARY OUTCOMES:
FGF23 peack or AUC | 12 hours
  We have chosen 24-72 hour AUC as our best predictionbased on limited previous data on this subject. Therefore, we will include other measurements of FGF23, namely the 12 hr peak and 12 hour AUC for FGF23 to analyze possible changes that occur prior to 24 hours.
Transtubular reabsorption of phosphate | 12 hours
  Renal phosphate transport is a complex interplay between freely filtered phosphate by the glomerulus, reabsorption of phosphate by brush border transporters in the proximal renal tubule, serum phosphate levels and hormonal regulation.
PTH | 12 hours
  We aim to explore if the postulated decreased 1,25 vitamin D leads to a secondary hyperparathyroidism leading to detrimental effects on bone. We hope to define this relationship further by investigating the timing and magnitude of changes in PTH over this short term study. The previous study by Rosenstock et al. 43 may have demonstrated initial increased in PTH that returned to a new baseline (data not available), but it should be noted that (1) the analysis presented is mean data and therefore some individuals likely have higher than average numbers, and (2) small changes in baseline PTH can have important changes in bone homeostasis over time.
1, 25 vitamin D | 12 hours
  In vivo and in vitro studies have demonstrated FGF23 is a potent regulator of 1 - hydroxylase causing rapid reductions in 1,25 vitamin D 66,74,75. Shimada et al. 66 demonstrated in rats that a single injection of FGF23 caused a rapid decrease in 1,25 vitamin D levels by 3 hours, prior to any changes in phosphate (9 hours) or PTH (no change). Therefore, we intend to define the extend and time course of change in 1,25 vitamin D in humans by SGLT2 inhibition.

CONTACTS AND LOCATIONS:
Overall Officials: Kelly B Roszko, M.D., Principal Investigator — National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

REFERENCES:
- [Derived] Blau JE, Bauman V, Conway EM, Piaggi P, Walter MF, Wright EC, Bernstein S, Courville AB, Collins MT, Rother KI, Taylor SI. Canagliflozin triggers the FGF23/1,25-dihydroxyvitamin D/PTH axis in healthy volunteers in a randomized crossover study. JCI Insight. 2018 Apr 19;3(8):e99123. doi: 10.1172/jci.insight.99123. eCollection 2018 Apr 19. PMID 29669938
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2014-DK-0195.html